CLINICAL TRIAL: NCT05582941
Title: Use of Human Blood Cells for the Identification of Early Biomarkers of Cognitive Damage
Brief Title: Biomarkers of Cognitive Impairment in Blood Cells
Acronym: COGNIMARK
Status: Completed | Type: Observational
Sponsor: University of the Balearic Islands (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Sponsor
Other Study IDs: IB 3799/18 PI
Record Dates: First submitted 2022-07-28; First posted 2022-10-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease; Dementia Due to Alzheimer's Disease (Disorder)
Keywords: Mild Cognitive Impairment; Alzheimer Disease; Blood cells; Adiposity; Nutrition
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples for analysis of gene expression and general clinical parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control: 20 individuals with no cognitive alterations or any other pathology which could alter cognitive performance or blood cells
  Interventions: Other: No intervention will be performed.
- Mild Cognitive Impairment Due to Alzheimer's Disease: MCI group: 20 individuals diagnosed with Mild Cognitive Impairment Due to Alzheimer's Disease with positive AD markers in cerebrospinal fluid
  Interventions: Other: No intervention will be performed.
- Dementia due to Alzheimer Disease: AD group: 20 individuals diagnosed with Dementia Due to Alzheimer Disease with positive AD markers in cerebrospinal fluid
  Interventions: Other: No intervention will be performed.

INTERVENTIONS:
Other: No intervention will be performed. — No intervention will be performed.

SUMMARY:
The aim of this study is to identify transcriptomic biomarkers in blood cells to diagnose early cognitive impairment. This would allow preventing the development of severe pathologies, such as Alzheimer Disease. In addition, this project will analyse the influence of adiposity, obesity, nutritional habits and physical activity on cognition.

DETAILED DESCRIPTION:
Blood cells constitute a minimally invasive material, which is presented as potentially suitable for addressing the identification of clinical diagnostic biomarkers. This study will compare gene expression in blood cells of patients with various degrees of cognitive alteration (mild cognitive impairment due to Alzheimer's disease and dementia due to Alzheimer's Disease) compared to control individuals, to identify early biomarkers of impaired cognition. The availability of non-invasive early biomarkers of cognitive dysfunction is highly relevant in the field of public health, from the point of view of being able to prevent or delay the onset and/or progression of dementia and other cognitive disorders. In addition, it is intended to establish the association between the biomarkers identified with nutritional imbalances and increased adiposity/obesity.

ELIGIBILITY:
1. Control group

   Inclusion criteria:
   * Age between 55-80 years
   * Absence of cognitive symptoms
   * Normal neuropsychological examination, (Clinical Dementia Rating, CDR = 0)

   Exclusion criteria:
   * Any disease that could influence their cognitive performance or blood cell parameters.
2. Group with Mild Cognitive Impairment Due to Alzheimer's Disease (MCI group)

   Inclusion criteria:
   * Age between 55-80 years
   * Established diagnosis of MCI
   * Cognitive deficit of 1.5 standard deviation in at least one of the neuropsychological tests performed, with no relevant functional repercussion (Functional Activities Questionnaire, FAQ<7 and CDR≤0.5)
3. Group with Dementia Due to Alzheimer Disease (AD)

Inclusion criteria:

* Age between 55-80 years
* Established diagnosis of Alzheimer's disease
* CDR ≥ 0.5 and positive AD markers in cerebrospinal fluid

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the participants are from Spain.
  * Control group: the majority are recruited from an Adult University (UOM, Universitat Oberta per Majors, University of the Balearic Island).
  * Mild Cognitive Impairment and Alzheimer Disease groups: are recruited from the University Hospital, Son Espases, Mallorca, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of semiquantitative gene expression of blood cells between the three groups | Baseline point (all groups)
  Gene expression analysis performed by real-time quantitative polymerase chain reaction (RT-qPCR). Percentage of semiquantitative gene expression between the groups: MCI vs Control, AD vs Control, and MCI vs AD
Mini-Mental State Examination (MMSE), questionnaire (numerical scale) | Baseline point (all groups)
  Cognitive test
Montreal Cognitive Assessment (MoCA), questionnaire (numerical scale) | Baseline point (all groups)
  Cognitive test
Cognitive Reserve Questionnaire (CRIq), questionnaire (numerical scale) | Baseline point (all groups)
  Cognitive test
Body composition (fat mass) | Baseline point (all groups)
  Percentage of fat mass measured using a dual energy x-ray absorptiometry (DXA) scanner

SECONDARY OUTCOMES:
Height (cm) | Baseline point (all groups)
  Basic anthropometric parameter, measured in centimeters with a tape-measure
Weight (kg) | Baseline point (all groups)
  Basic anthropometric parameter, measured using a scale
Waist-hip ratio (numerical ratio) | Baseline point (all groups)
  Basic anthropometric parameter. Waist circumference (cm) and hip circumference (cm) will be combined to report waist-hip ratio (waist(cm)/hip(cm))
Blood pressure (mm Hg) | Baseline point (all groups)
  Basic anthropometric parameter, measured in millimeters of mercury with a blood pressure monitor
Body Mass Index (BMI) (kg/m2) | Baseline point (all groups)
  Basic anthropometric parameter. Weight and height will be combined to report BMI in kg/m^2
Complete blood count test (numbers of cells/mcL) | Baseline point (all groups)
  Circulating parameter (from blood sample). It will be measured: red blood cells, white blood cells (neutrophils, lymphocytes, monocytes, eosinophils, basophils) and platelets. All of them measured in numbers of cells/mcL by a complete blood count test.
Plasma glucose (mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Triglycerides (TG, mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Total cholesterol (mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
High-density lipoprotein cholesterol (HDL-C,mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Low-density lipoprotein cholesterol (LDL-C, mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Aspartate aminotransferase (AST, U/L) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Alanine aminotransferase (ALT, U/L) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Gamma-glutamyl transpeptidase (GGT, U/L) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Transpeptidase (GGT, U/L) | Baseline point (all groups)
  Circulating parameter (from blood sample)
C-reactive protein (CRP, mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Apolipoprotein E (APOE, mg/dL) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Glycated hemoglobin (HbA1c, %) | Baseline point (all groups)
  Circulating parameter (from blood sample)
Test on nutritional habits, questionnaire (numerical scale) | Baseline point (all groups)
  Lifestyle test. Test on nutritional habits based on a 14-item Mediterranean diet questionnaire
International Physical Activity Questionnaire, IPAQ (numerical scale) | Baseline point (all groups)
  Lifestyle test, specifically a physical activity test
STOP-BANG Sleep Apnea Questionnaire (numerical scale) | Baseline point (all groups)
  Lifestyle test, specifically a screening for obstructive sleep apnea in adults
Gait Speed Test (m/s) | Baseline point (all groups)
  Gait speed is recorded on a 4 meter walkway with 2 meter non-instrumented walkway segments at each end to allow for acceleration and deceleration. Gait speed recorded is the average of the speed for the two trials

CONTACTS AND LOCATIONS:
Overall Officials: Paula Oliver, Professor, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma, Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will be shared in due time if considered relevant for other research. With our current objectives, it is not considered necessary.

REFERENCES:
- See also: Article from the research group that supports the relation between normal-weight obesity in rodents and cognitive impairment in rats. — http://pubmed.ncbi.nlm.nih.gov/29566703/